CLINICAL TRIAL: NCT00786656
Title: NCI Community Cancer Center Pilot Program Patient Survey
Brief Title: Community Cancer Centers Pilot Patient Survey
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999909026; 09-C-N026
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2015-05-11

CONDITIONS: Malignant Neoplasms; Cancer
Keywords: Navigation; Coordination; Cancer Care; Patient Experience; Cancer; Patient Survey
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

SUMMARY:
Background:

* Studies suggest that cancer patients diagnosed and treated in a facility with multi-specialty care and clinical research may live longer and have a better quality of life than patients treated elsewhere.
* The NCI Community Cancer Centers Pilot Program (NCCCP) is a 3-year program to test the concept of a national network of community cancer centers to expand cancer research and deliver the most advanced cancer care to Americans in their own communities.
* The pilot program includes a survey of cancer patients receiving care at the pilot sites.

Objectives:

* To gain an understanding of the experiences of adult patients who receive services at the NCCCP pilot sites and assess if and how their experience changes over the study period. Data about the following are collected:
* Patients information needs and awareness of the NCCCP program
* Clinical trials experience
* Access to health care
* Perspectives on patient-provider communication
* Experiences with patient navigation, self-management, medical decision-making and survivorship
* Satisfaction with care and quality of life

Eligibility:

* Patients 21 years or older at the time of diagnosis
* Treatment at the cancer center for at least 3 months since July 1, 2007

Design:

* Participants complete a 25-minute questionnaire covering the care they received at their cancer center, their experience with making medical appointments and how long they waited to see the doctor. The survey includes information on the following:
* Services at the cancer center
* Getting needed care
* Assistance for patients and their families
* Communication with the cancer care team
* Clinical trials
* Care after finishing treatment
* Evaluation of care
* Health and medical history
* Background information (demographics)

DETAILED DESCRIPTION:
BACKGROUND:

The NCI Community Cancer Centers Pilot Program (NCCCP), http://ncccp.cancer.gov, is a three-year pilot program to test the concept of a national network of community cancer centers to expand cancer research and deliver the latest, most advanced cancer care to a greater number of Americans in the communities in which they live.The pilot program is designed to encourage the collaboration of private-practice medical, surgical, and radiation oncologists, with close links to NCI research and to the network of 63 NCI-designated cancer Centers principally based at large research universities. NCI contracted with RTI International (ww.rti.org) to conduct a comprehensive evaluation of the NCCCP pilot program using multiple methodologies, including a survey of cancer patients receiving care at the pilot sites.

OBJECTIVES:

The goal of the patient survey is to gain an understanding of the clinical experiences of adult patients who receive services at the NCCCP pilot sites and to assess if and how their experience change over the pilot period. Specifically, the survey instrument seeks to collect data about patients information needs and awareness of the NCCCP program; clinical trials experience; access to health care; perspectives on patient-provider communication; and experiences with patient navigation, self-management, medical decision making, and survivorship; as well as their satisfaction with care and quality of life.

ELIGIBILITY:

Each of the ten participating Centers will create a de-identified electronic file of all patients who meet the inclusion criteria:

1. living patients who are listed on a NCCCP site s cancer registry;
2. cancer patients age 21 years and older at the time of sampling; and
3. cancer patients who had 1or more cancer treatment outpatient visits at their Cancer Center since July 1, 2007 for the 1st round of data collection, and since July 1, 2009 for the second data collection. Center will create this file using their cancer registry and assign each individual a unique identification (ID) number.

DESIGN:

Each file containing the universe of eligible patients will be sent to RTI, from which 475 patients from each Center s list will be randomly selected. RTI will send a list back to each Center indicating which 475 patient IDs were selected for inclusion in the survey. The Center staff will match selected patient back to their master list using the Study ID number to identify patients included in the survey. RTI will deliver 475 pre-paid patient survey packets to each Center. The packets will include all required items except a Patient Notification Letter, which is a cover letter introducing the study and provides instructions on how to complete the survey. To protect patient privacy, Center staff will be responsible for generating the mailing labels and personalized Patient Notification Letter, and mailing the packets.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Living patients who are listed on an NCCCP site s cancer registry
* Cancer patients age 21 years and older at the time of sampling
* Cancer patients who had 1 or more cancer treatment outpatient visits at their cancer center since July 1, 2007 for the first survey round and since July 1, 2009 for the second round of the survey.

EXCLUSION CRITERIA:

* Persons under the age of 21 at the time of sampling.
* Persons not in the cancer registry
* Cancer patients without at least 1 or more cancer treatment outpatient visits since July 1, 2007 for the first survey round and since July 1, 2009 for the second round of the survey.
* Cancer patients who are deceased at the time of sampling

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3955 (Actual)
Dates: Start 2008-11-03; Study Completion 2015-05-11

PRIMARY OUTCOMES:
Evaluation of NCCCP Pilot Program

SECONDARY OUTCOMES:
Gain an understanding of the patients' perspective on the NCCCP Pilot Program and to assess how well health care and informational needs are being met.

CONTACTS AND LOCATIONS:
Overall Officials: Irene P Prabhu Das, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Research Triangle Institute International, Research Triangle Park, North Carolina, United States